CLINICAL TRIAL: NCT07062120
Title: Efficacy and Safety of 30% Salicylic Acid and 10% Nicotinamide Combined Therapy in Melasma: A Randomized Placebo Controlled Study
Brief Title: Efficacy and Safety of 30% Salicylic Acid and 10% Nicotinamide Combined Therapy in Melasma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Second Affiliated Hospital of Xi'an Jiaotong University (Other)
Responsible Party: Principal Investigator, Weihui Zeng, Professor, Second Affiliated Hospital of Xi'an Jiaotong University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2021016
Record Dates: First submitted 2025-06-29; First posted 2025-07-14 (Actual); Last update posted 2025-07-14 (Actual); Status verified 2025-07

CONDITIONS: Melasma
Keywords: Melasma; salicylic acid; nicotinamide; chemical peeling
MeSH Terms: conditions — Melanosis

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- 30% SSA group(SSA) (Experimental): 30% SSA treatment were with 2-week intervals for eight sessions, and the follow-up was conducted 2 weeks after the last session
  Interventions: Other: Supramolecular salicylic acid(SSA) (30%); Other: Nicotinamide simulator
- 10% NAM group(NAM) (Experimental): 10% NAM treatment were twice a day during the entire follow-up period
  Interventions: Other: Nicotinamide(NAM)(10%); Other: Supramolecular salicylic acid simulator
- 30% SSA plus 10% NAM group (SSA+NAM) (Experimental): 30% SSA treatment were with 2-week intervals for eight sessions, and 10% NAM treatment were twice a day during the entire follow-up period
  Interventions: Other: Nicotinamide(NAM)(10%); Other: Supramolecular salicylic acid(SSA) (30%)
- Placebo control group (Ctrl) (Placebo Comparator): received the same course of treatment in the same dosage form that does not contain SA and NAM.
  Interventions: Other: Supramolecular salicylic acid simulator; Other: Nicotinamide simulator

INTERVENTIONS:
Other: Nicotinamide(NAM)(10%) — The active niacinamide form of vitamin B3, NAM is routinely employed as a pigmentation-reducing agent in melasma treatment protocols
  Arms: 10% NAM group(NAM); 30% SSA plus 10% NAM group (SSA+NAM)
Other: Supramolecular salicylic acid(SSA) (30%) — Salicylic acid, a superficial chemical peel, has been widely used in treating melasma. Breakthroughs in supramolecular design have addressed its irritancy profile through engineered SA complexes with improved water dispersibility
  Arms: 30% SSA group(SSA); 30% SSA plus 10% NAM group (SSA+NAM)
Other: Supramolecular salicylic acid simulator — the same course of treatment in the same dosage form that does not contain salicylic acid
  Arms: 10% NAM group(NAM); Placebo control group (Ctrl)
Other: Nicotinamide simulator — the same course of treatment in the same dosage form that does not contain nicotinamide
  Arms: 30% SSA group(SSA); Placebo control group (Ctrl)

SUMMARY:
This prospective, randomized, placebo-controlled study evaluated the synergistic effects of 30% salicylic acid (SA) chemical peels and topical 10% nicotinamide (NAM) in 56 patients with moderate-to-severe melasma. Participants were divided into four groups: placebo control, SA peels alone (every 2 weeks for 8 sessions), NAM cream alone (twice daily for 16 weeks), and combination therapy (SA+NAM). The investigators investigated the efficacy and safety of 30%SA chemical peeling combined with 10% NAM.

DETAILED DESCRIPTION:
Background:Melasma is a common skin disease manifested as brown patches with symmetrical distribution and irregular boundaries. Chemical peeling with salicylic acid (SA) is widely used in the treatment of melasma. Nicotinamide (NAM) is a common whitening agent and has a good effect in the treatment of melasma. In the present study, the investigators investigated the efficacy and safety of 30%SA chemical peeling combined with 10% NAM.

Methods: 56 moderate-to-severe melasma patients were enrolled and randomly assigned into the control group, SA group, NAM group, and SA+NAM group. SA treatment was given at an interval of 2 weeks for 8 treatment sessions (week 0, 2, 4, 6, 8, 10, 12, 14). NAM was applied twice a day for 16w. Photos, mMASI score, and skin indices (TEWL, skin hydration, melanin index, erythema index, red areas score, and UV spots score) were assessed at 0, 2, 4, 6, 8,10,12, and 14 weeks. Side effects, efficacy and satisfactory scores were recorded.

Limitations: Retrospective single-center design and small sample size.

ELIGIBILITY:
Inclusion Criteria:

1. Males and nonpregnant females, aged 18-60 years old;
2. Diagnosed with melasma;
3. Patients with good cognitive function and normal mental status;
4. Patients with good communication skills;
5. Voluntary participation in the study and signing of informed consent form.

Exclusion Criteria:

1. pregnancy or lactation;
2. pigmentation from other causes, such as hormonal dermatitis, cosmetic dermatitis, etc;
3. established allergy to SA or NAM;
4. active skin infection;
5. systemic diseases, such as immunodeficiency disease, diabetes, lupus erythematosus, etc;
6. having facial surgery, laser treatment, or whitening products in the past three months;
7. neurological or psychiatric disorders.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2021-04-01 (Actual); Study Completion 2021-04-01 (Actual)

PRIMARY OUTCOMES:
mMASI score | From enrollment to week 16
  The Primary outcomes were pre-defined as mMASI score and percent change in mMASI score, which was calculated as (mMASI at baseline-mMASI after treatment)/ mMASI at baseline × 100% and was graded as recovery (≥90%), obvious improvement (60-89%), improvement (20-59%), and no improvement (<20%).

SECONDARY OUTCOMES:
melanin index | From enrollment to week 16
  Use non-invasive skin analyzer to measure the melanin index on the patient's facial skin at each follow-up visit.
The skin hydration | From enrollment to week 16
  Use non-invasive skin analyzer to measure the skin hydration on the patient's facial skin at each follow-up visit.
transepidermal water loss | From enrollment to week 16
  Use non-invasive skin analyzer to measure the transepidermal water loss on the patient's facial skin at each follow-up visit.
erythema index | From enrollment to week 16
  Use non-invasive skin analyzer to measure the erythema index on the patient's facial skin at each follow-up visit.
Actinic damage (UV spots) | From enrollment to week 16
  Use VISIA to measure the UV spots on the patient's facial skin at each follow-up visit.
patient satisfaction evaluation | week 16
  Patient satisfaction was evaluated as very satisfied, satisfied, relatively satisfied and dissatisfied.

CONTACTS AND LOCATIONS:
Overall Officials: Weihui Zeng, Study Chair — Second Affiliated Hospital of Xi'an Jiaotong University
Locations (1):
- The Second Affiliated Hospital of Xi'an Jiaotong Universi, Xi'an, Shaanxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Fania L, Mazzanti C, Campione E, Candi E, Abeni D, Dellambra E. Role of Nicotinamide in Genomic Stability and Skin Cancer Chemoprevention. Int J Mol Sci. 2019 Nov 26;20(23):5946. doi: 10.3390/ijms20235946. PMID 31779194
- [Background] Madaan P, Sikka P, Malik DS. Cosmeceutical Aptitudes of Niacinamide: A Review. Recent Adv Antiinfect Drug Discov. 2021;16(3):196-208. doi: 10.2174/2772434416666211129105629. PMID 34844552
- [Background] Searle T, Al-Niaimi F, Ali FR. The top 10 cosmeceuticals for facial hyperpigmentation. Dermatol Ther. 2020 Nov;33(6):e14095. doi: 10.1111/dth.14095. Epub 2020 Sep 4. PMID 32720446
- [Background] Spierings NMK. Melasma: A critical analysis of clinical trials investigating treatment modalities published in the past 10 years. J Cosmet Dermatol. 2020 Jun;19(6):1284-1289. doi: 10.1111/jocd.13182. Epub 2019 Oct 11. PMID 31603285
- [Background] McKesey J, Tovar-Garza A, Pandya AG. Melasma Treatment: An Evidence-Based Review. Am J Clin Dermatol. 2020 Apr;21(2):173-225. doi: 10.1007/s40257-019-00488-w. PMID 31802394
- [Background] Kwon SH, Na JI, Choi JY, Park KC. Melasma: Updates and perspectives. Exp Dermatol. 2019 Jun;28(6):704-708. doi: 10.1111/exd.13844. Epub 2018 Dec 21. PMID 30422338
- [Background] Ogbechie-Godec OA, Elbuluk N. Melasma: an Up-to-Date Comprehensive Review. Dermatol Ther (Heidelb). 2017 Sep;7(3):305-318. doi: 10.1007/s13555-017-0194-1. Epub 2017 Jul 19. PMID 28726212